CLINICAL TRIAL: NCT06086275
Title: Oral Buprenorphine as a Novel Low-Dose Induction Strategy for Individuals With Opioid Use Disorder
Brief Title: Oral Buprenorphine as a Novel Low-dose Induction Strategy for Opioid Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2023P002634
Record Dates: First submitted 2023-10-03; First posted 2023-10-17 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: All participants will first receive the IV arm in fixed order, in an open-label fashion. Subsequently, participants will be randomized to the two PO.
Masking Description: All portions will be open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 8mg PO buprenorphine (Experimental): After the open-label period, the participant will receive 8mg PO, then 16mg PO will be administered in the following visit.
  Interventions: Drug: Buprenorphine
- 16mg PO buprenorphine (Experimental): After the open-label period, the participant will receive 16mg PO, then 8mg PO will be administered in the following visit.
  Interventions: Drug: Buprenorphine
- 0.15mg IV Dose (Experimental): The first dose administered will be fixed to an open-label 0.15mg IV dose.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — At each visit, the participant will receive a single dose of buprenorphine, either 0.15mg IV, 8mg PO, or 16mg PO. The order for the first dose administered will be fixed to the IV dose, and the subsequent doses will be randomized and counterbalanced to 8mg or 16mg PO.

SUMMARY:
This is a human laboratory-based, randomized, cross-over study in which buprenorphine will be administered to healthy volunteers (n=22) in 3 separate inpatient 2-night visits, at least 1 week apart. At each visit, the participant will receive a single dose buprenorphine, either 0.15mg IV, 8mg PO, or 16mg PO. The order for the first dose administered will be fixed to the IV dose, and the subsequent doses will be randomized and counterbalanced to 8mg or 16mg PO. Participants will be given naltrexone to produce opioid blockade to eliminate the risk for opioid dependence in individuals without OUD. Timed blood samples will be collected up to 24 hours.

DETAILED DESCRIPTION:
The approach is to conduct a randomized, cross-over trial in a controlled human laboratory setting with healthy volunteers (n=22). After obtaining informed consent, eligible participants will be scheduled for 3 separate two-night test days to receive 0.15mg IV, 8mg PO, or 16mg PO of buprenorphine. The first dose administered will be fixed to an open-label IV dose, and the subsequent doses will be randomized and counterbalanced to 8mg or 16mg PO. Visits will be scheduled at least 1 week apart to allow for washout of drug. One hour prior to receipt of the buprenorphine dose, all participants will be fed a standardized light breakfast. The IV dose will be given after establishing IV access, while the PO doses will be swallowed whole. Participants will also receive oral naltrexone 100mg 24 hours prior to each dosing to provide blockade at the mu-receptor, as well as 50mg PO at the study visit itself prior to receipt of buprenorphine. Timed blood samples will be collected in heparinized Vacutainer tubes via a catheter in the antecubital vein at baseline, and at 0.5, 1, 2, 4, 8, and 24 hours. Samples will be centrifuged and frozen until analysis.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults aged 18 and above.
* In good physical health as determined by routine medical screening consisting of a complete physical exam, safety labs and EKG.
* Baseline vital signs with HR between 60 and 100, SBP between 90 and 160mmHg, and respiratory rate between 12 and 20 breaths per minute.
* Prior personal history of opioid use, therapeutic or non-therapeutic in past the 12 months.

Exclusion Criteria:

* DSM-5 diagnosis of any substance use disorder excluding tobacco.
* Presence of any alcohol, cannabis, opioids (including methadone, buprenorphine) or any other illicit substances on urine toxicology at any study visit, including cocaine, amphetamines, and benzodiazepines.
* Receiving treatment with opioid analgesic in last 60 days, or anticipate requiring opioids during the proposed trial, or up to 30 days after the trial completion
* Baseline PHQ-9 or GAD7 > 10 (i.e. moderate depression/anxiety)
* History of chronic pain
* Psychotic disorder, active suicidality or homicidally, or any psychiatric condition that impair ability to provide informed consent.
* History of hypersensitivity or allergy to buprenorphine or naltrexone
* Pregnant or breastfeeding.
* Liver function test greater than 3 times upper normal limit.
* Receiving medications that are strong or moderate CYP34A inducers or inhibitors (including but not limited to ketoconazole, itraconazole, clarithromycin, fluconazole, erythromycin), in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Plasma-Concentration Curves (AUC) of Buprenorphine | Baseline, 0.5, 1, 2, 4, 8, and 24 hours after study drug administration.
  The area under the plasma concentration curves (AUC) of buprenorphine will be determined. Timed blood samples will be collected in heparinized Vacutainer tubes via a catheter in the antecubital vein at baseline, and at 0.5, 1, 2, 4, 8, and 24 hours. Samples will be centrifuged and frozen until analysis.

SECONDARY OUTCOMES:
Maximum Plasma Concentration | Baseline, 0.5, 1, 2, 4, 8, and 24 hours after study drug administration.
  Plasma data will be used to calculate maximum plasma concentration (Cmax) for buprenorphine, norbuprenorphine, and their glucuronides.
Time to Maximum Plasma Concentration | Baseline, 0.5, 1, 2, 4, 8, and 24 hours after study drug administration.
  Plasma data will be used to calculate time to maximum plasma concentration (Tmax) for buprenorphine, norbuprenorphine, and their glucuronides.
Volume of Distribution | Baseline, 0.5, 1, 2, 4, 8, and 24 hours after study drug administration.
  Plasma data will be used to calculate volume of distribution (Vd) for buprenorphine, norbuprenorphine, and their glucuronides.
Elimination half-life | Baseline, 0.5, 1, 2, 4, 8, and 24 hours after study drug administration.
  Plasma data will be used to calculate elimination half-life (t1/2) for buprenorphine, norbuprenorphine, and their glucuronides.
Total Clearance | Baseline, 0.5, 1, 2, 4, 8, and 24 hours after study drug administration.
  Plasma data will be used to calculate total clearance (CL) for buprenorphine, norbuprenorphine, and their glucuronides.
Pupil Size | Baseline, 0.5, 1, 2, 4, 8, and 24 hours after study drug administration.
  Pupil size will be measured through visual inspection both before and after buprenorphine dosing to confirm opioid blockade.
The Drug Effects Questionnaire | Baseline, 0.5, 1, 2, 4, 8, and 24 hours after study drug administration.
  To confirm opioid blockade, subjective and objective opioid effects will be measured using previously validated Drug Evaluation Questionnaire (DEQ). The DEQ is a 5-item questionnaire where participants answer questions on a sliding scale from 0-100, where 0 indicates lower levels drug effects and 100 indicates higher levels of drug effects.
Buccal Swab | will be done once at the baseline visit.
  DNA testing to check 3A4 activity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's hospital, Boston, Massachusetts, United States